CLINICAL TRIAL: NCT03278457
Title: Risk Stratification Using Positron Emission Tomography (PET) in Hypertrophic Cardiomyopathy (HCM)
Brief Title: Risk Stratification Using PET in HCM
Acronym: HCM-PET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Gävleborg (Other)
Collaborators: Landstinget i Värmland (Other); Dalarna County Council, Sweden (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017021
Record Dates: First submitted 2017-08-21; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; implantable cardioverter defibrillator; positron emission tomography
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography — Positron Emission Tomography

SUMMARY:
The overall rationale is to reduce the risk of sudden cardiac death in individuals with hypertrophic cardiomyopathy (HCM). The novel approach of this study is to correlate Positron Emission Tomography (PET) findings to ventricular arrhythmias detected by the implantable cardioverter defibrillator (ICD). This could potentially lead to an improved risk stratification of HCM patients.

DETAILED DESCRIPTION:
Positron Emission Tomography (PET) is a functional imaging technique that utilizes radioactive tracers to gain information on physiological or pathophysiological processes in vivo. Different tracers can provide information on different processes of interest. In cardiology, metabolic processes consuming oxygen (aerobic) can be studied with 11-Carbon-Acetate, sympathetic innervation can be studied with 11-Carbon-hydroxyephedrine and using 15-Oxygen-water the myocardial blood flow. Structural information of the heart such as left ventricular mass, left ventricular volumes and wall thickness can also be calculated with PET.

The aim is to correlate PET parameters and burden of ventricular arrhythmias in order to improve risk stratification in HCM.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic cardiomyopathy, implantable cardioverter defibrillator, informed consent

Exclusion Criteria:

* Patients younger than 18 years, pregnancy, breast feeding, claustrophobia, intolerance/allergic reaction to adenosin or mannitol, severe hypotension, unstable angina pectoris, incompensated systolic heart failure, increased intracranial pressure, hypovolemia, dipyramidole.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with hypertrophic cardiomyopathy (HCM) and an implantable defibrillator (ICD)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-01-03 (Estimated); Study Completion 2018-06-03 (Estimated)

PRIMARY OUTCOMES:
Ventricular tachycardia (VT) vs myocardial blood flow | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter Myocardial blood flow (MBF)
Ventricular tachycardia (VT) vs ejection fraction | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter ejection fraction (EF)
Ventricular tachycardia (VT) vs mass | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter mass
Ventricular tachycardia (VT) vs wall thickness | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter wall thickness
Ventricular tachycardia (VT) vs oxygen consumption | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter oxygen consumption (MVO2)
Ventricular tachycardia (VT) vs sympathetic innervation | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter sympathetic innervation (retention index)
Ventricular tachycardia (VT) vs myocardial external efficiency | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter myocardial external efficiency (MEE)
Ventricular tachycardia (VT) vs stroke work | History of VT since receiving an implantable defibrillator within last 15 years
  Ventricular tachycardia vs positron emissions tomography parameter stroke work (SW)

SECONDARY OUTCOMES:
Atrial fibrillation (AF) vs myocardial blood flow | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter myocardial blood flow
Atrial fibrillation (AF) vs ejection fraction | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter ejection fraction (EF)
Atrial fibrillation (AF) vs mass | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter mass
Atrial fibrillation (AF) vs wall thickness | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter wall thickness
Atrial fibrillation (AF) vs oxygen consumption | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter oxygen consumption (MVO2)
Atrial fibrillation (AF) vs sympathetic innervation | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter sympathetic innervation (retention index)
Atrial fibrillation (AF) vs myocardial external efficiency | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter myocardial external efficiency (MEE)
Atrial fibrillation (AF) vs stroke work | History of VT since receiving an implantable defibrillator within last 15 years
  Atrial fibrillation vs positron emissions tomography parameter stroke work (SW)
Atrial size vs ventricular tachycardia | History of VT since receiving an implantable defibrillator within last 15 years
  atrial diameter, volume vs ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sörensen, MD PhD, Principal Investigator — Region Gävleborg
Locations (1):
- Region Gavleborg, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Authors/Task Force members; Elliott PM, Anastasakis A, Borger MA, Borggrefe M, Cecchi F, Charron P, Hagege AA, Lafont A, Limongelli G, Mahrholdt H, McKenna WJ, Mogensen J, Nihoyannopoulos P, Nistri S, Pieper PG, Pieske B, Rapezzi C, Rutten FH, Tillmanns C, Watkins H. 2014 ESC Guidelines on diagnosis and management of hypertrophic cardiomyopathy: the Task Force for the Diagnosis and Management of Hypertrophic Cardiomyopathy of the European Society of Cardiology (ESC). Eur Heart J. 2014 Oct 14;35(39):2733-79. doi: 10.1093/eurheartj/ehu284. Epub 2014 Aug 29. No abstract available. PMID 25173338
- [Background] Maron BJ, Olivotto I, Spirito P, Casey SA, Bellone P, Gohman TE, Graham KJ, Burton DA, Cecchi F. Epidemiology of hypertrophic cardiomyopathy-related death: revisited in a large non-referral-based patient population. Circulation. 2000 Aug 22;102(8):858-64. doi: 10.1161/01.cir.102.8.858. PMID 10952953
- [Background] Timmer SA, Germans T, Gotte MJ, Russel IK, Dijkmans PA, Lubberink M, ten Berg JM, ten Cate FJ, Lammertsma AA, Knaapen P, van Rossum AC. Determinants of myocardial energetics and efficiency in symptomatic hypertrophic cardiomyopathy. Eur J Nucl Med Mol Imaging. 2010 Apr;37(4):779-88. doi: 10.1007/s00259-009-1350-3. Epub 2010 Jan 13. PMID 20069294
- [Background] Kofflard MJ, Ten Cate FJ, van der Lee C, van Domburg RT. Hypertrophic cardiomyopathy in a large community-based population: clinical outcome and identification of risk factors for sudden cardiac death and clinical deterioration. J Am Coll Cardiol. 2003 Mar 19;41(6):987-93. doi: 10.1016/s0735-1097(02)03004-8. PMID 12651046
- [Background] Timmer SA, Germans T, Gotte MJ, Russel IK, Lubberink M, Ten Berg JM, Ten Cate FJ, Lammertsma AA, Knaapen P, van Rossum AC. Relation of coronary microvascular dysfunction in hypertrophic cardiomyopathy to contractile dysfunction independent from myocardial injury. Am J Cardiol. 2011 May 15;107(10):1522-8. doi: 10.1016/j.amjcard.2011.01.029. Epub 2011 Mar 4. PMID 21377644